CLINICAL TRIAL: NCT05710289
Title: A Prospective Blood Collection Study to Assess the Immunogenicity of Homologous Booster Combinations of COVID-19 Vaccines Available Under Emergency Use Authorization Among Adults of 18 Years and Older.
Brief Title: A Blood Collection Study to Assess the Immunogenicity of Nationally Authorized Homologous COVID-19 Booster Vaccines Among Adult Vaccinees.
Status: Withdrawn | Type: Observational
Why Stopped: Sponsor's decision
Sponsor: SK Bioscience Co., Ltd. (Industry)
Collaborators: International Vaccine Institute (Other)
Responsible Party: Sponsor
Other Study IDs: GBP510_005
Record Dates: First submitted 2023-01-30; First posted 2023-02-02 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Immunity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Primary series of mRNA-1273: Manufactured by ModernaTX
  Interventions: Biological: Immune Responses
- Primary series of ChAdOx1 nCOV-19: Manufactured by Astrazeneca or Serum Institute of India Pvt., Ltd
  Interventions: Biological: Immune Responses
- A single dose vaccination of Ad26.COV2.S: Manufactured by Janssen Pharmaceuticals/Johnson & Johnson
  Interventions: Biological: Immune Responses
- Primary series of BNT162b2: Manufactured by Pfizer
  Interventions: Biological: Immune Responses
- Primary series of BBIBP-CorV: Manufactured by Sinopharm
  Interventions: Biological: Immune Responses
- Primary series of CoronaVac: Manufactured by Sinovac
  Interventions: Biological: Immune Responses

INTERVENTIONS:
Biological: Immune Responses — To compare the immune responses against the original strain and circulating strain prior to and post homologous dose of WHO EUA qualified COVID-19 vaccine in adults aged 18 years and older regardless of prior history of SARS-CoV-2 infection with immunogenicity profile of single heterologous dose by GBP510 vaccine acquired from GBP510_004 study.

SUMMARY:
The purpose of this study is to assess the immunogenicity of nationally available pre-defined homologous booster vaccination of a SARS-CoV-2 WHO EUA qualified vaccination in adults aged 18 years and older

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 18 years of age and older, at the time of signing the informed consent.
* Participants who are healthy or medically stable as determined by medical evaluation including medical history, physical examination, and medical judgement of the investigator.
* Participants who are able to attend all scheduled visits and comply with all study procedures.
* Participants who received primary vaccination of 1 of 6 different WHO EUA qualified COVID-19 vaccine (mRNA-1273, ChAdOx1 nCOV-19, Ad26.COV2.S, BNT162b2, BBIBP-CorV, CoronaVac) at least 12 weeks of gap prior to first homologous booster vaccination and with no history of other COVID-19 vaccination, including booster doses.
* Participants who complete a qualitative test for antibody to SARS-CoV-2 nucleocapsid proteins at screening for assessment of previous SARS-CoV-2 infection.
* Female participants with a negative urine or serum pregnancy test at screening.
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.

Exclusion Criteria:

* Concurrent or past SARS-CoV-2 infection within 12 weeks prior to the booster study vaccination confirmed by virological or serological testing .
* History of congenital, hereditary, acquired immunodeficiency, or autoimmune disease.
* History of bleeding disorder or thrombocytopenia which is contraindicating to take blood sample.
* History of malignancy within 1 year prior to the screening (with the exception of malignancy with minimal risk of recurrence at the discretion of the investigator).
* Significant unstable chronic or acute illness that, in the opinion of the investigator, might pose a health risk to the participant if enrolled, or could interfere with the protocol-specified activities, or interpretation of study results.
* Any other conditions which, in the opinion of the investigator, might interfere with the evaluation of the study objectives (e.g., alcohol or drug abuse, neurologic or psychiatric conditions).
* Receipt of any medications or vaccinations intended to prevent COVID-19 except for the pre-defined COVID-19 vaccines expected to be given prior to screening (mRNA-1273, ChAdOx1 nCOV-19, Ad26.COV2.S, BNT162b2, BBIBP-CorV, CoronaVac).
* Receipt of any vaccine within 4 weeks prior to the booster vaccination or planned receipt of any vaccine from enrollment through 4 weeks after the booster vaccination, except for influenza vaccination, which may be received at least 2 weeks prior to the booster vaccination.
* Receipt of immunoglobulins and/or any blood or blood products within 12 weeks prior to the booster vaccination.
* Chronic use (more than 2 consecutive weeks) of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy; or long-term systemic corticosteroid therapy (≥10mg prednisone/day or equivalent for more than 2 consecutive weeks) within 12 weeks prior to the booster vaccination. The use of topical and nasal glucocorticoids will be permitted.
* Participation in another clinical study and or concurrent, planned participation in another clinical study with study intervention during the study period.
* Investigators, or study staff who are directly involved in the conduct of this study or supervised by the investigator, and their respective family members.
* Donation of ≥450mL of blood product within 4 weeks prior to screening, or planned donation of blood product during the study period

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Available WHO EUA qualified homologous booster vaccination against SARS-Cov-2 among adults 18 Years and older participants, regardless of past SARS-CoV-2 infection history confirmed by either serological or virological test method at baseline.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-02 (Estimated); Primary Completion 2024-02 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
GMT of neutralizing antibody to SARS-CoV-2 | Through study completion, an average of 1 year
  Measured by wild-type virus neutralization assay
GMFR and percentage of participants with ≥4-fold rise of neutralizing antibody to SARS-CoV-2 | Through study completion, an average of 1 year
  Measured by Wild-type virus neutralization assay
GMT of SARS-CoV-2 RBD-binding IgG antibody | Through study completion, an average of 1 year
  Measured by ELISA
GMFR and percentage of participants with ≥4-fold rise of SARS-CoV-2 RBD-binding IgG antibody | From baseline (Visit 1) to each subsequent time point.
  Measured by ELISA
Cell-mediated response for both Th1 and Th2 cytokines | through study completion, an average of 1 year (Visit 1,3,6 and 7)
  Measured by ELISpot and/or FluoroSpot, and for both CD4+ and CD8+ T-cells measured by FACS

CONTACTS AND LOCATIONS:
Overall Officials: Santa K Das, MD, Principal Investigator — Study Principal Investigator

IPD SHARING:
Plan to Share IPD: No